CLINICAL TRIAL: NCT06499415
Title: Combination Therapy of 5-Fluorouracil and CALcipotriol Versus 5-Fluorouracil in the Treatment of Actinic Keratosis: a Multicentre Randomized Controlled Clinical Trial
Brief Title: Combination Therapy of 5-Fluorouracil and CALcipotriol Versus 5-Fluorouracil in the Treatment of Actinic Keratosis
Acronym: CALM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-511409-42-00
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Actinic Keratoses
Keywords: 5-Fluorouracil; Calcipotriol
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator, who is also a physician and will evaluate treatment effect, is blinded to the allocated treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- topical 5FU-CAL, twice daily, during 4 or 6 consecutive days (Experimental): Treatment duration is based on treatment location
  Interventions: Drug: 5FU-Calcipotriol
- topical 5FU, twice daily, 7 days a week, during 4 weeks (Active Comparator)
  Interventions: Drug: 5-FU 50 MG/ML Topical Cream

INTERVENTIONS:
Drug: 5FU-Calcipotriol — topical 5FU-CAL, twice daily, during 4 or 6 consecutive days, depending on the treatment location
  Arms: topical 5FU-CAL, twice daily, during 4 or 6 consecutive days
Drug: 5-FU 50 MG/ML Topical Cream — topical 5FU, twice daily, 7 days a week, during 4 weeks
  Arms: topical 5FU, twice daily, 7 days a week, during 4 weeks

SUMMARY:
5-Fluorouracil (5FU) is proven to be the most effective therapy in field directed treatment for AK, with Jansen et al. reporting a 1-year probability of treatment success of 74.7%. However, treatment with 5FU is associated with side effects, like erythema, itching, a burning sensation and crusting, and a burdensome dosing regimen of twice daily application for four weeks. This long treatment duration in combination with side-effects and overall lifestyle adjustments during treatment can be the reason for poor adherence and premature termination, and it can also lead to future refusal of 5FU therapy. Therefore, room for improvement lies in increasing the tolerability, in terms of side effects or treatment duration, while maintaining the efficacy of 5FU in the treatment of AK.

Addition therapy, which can shorten the duration of treatment, might be the key to success. Calcipotriol (CAL) enhances thymic stromal lymphopoietin (TSLP), an epithelium-derived cytokine, which promotes antitumor immunity. Therefore, it is known to have a synergistic effect when combined with 5FU in the treatment of AK. This suggests that short-term treatment with 5FU-CAL is effective and provides the opportunity to shorten duration of treatment, thereby improving tolerability of treatment and full adherence to the treatment regimen.

However, no study compared 5FU-CAL combination therapy with standard 5FU treatment for a duration of 28 days. This study aims to evaluate whether a short course of combination therapy with 5FU-CAL is non-inferior to a full course of 5FU monotherapy with respect to the 1-year probability of treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Adults above 18 years of age
* Clinical and dermoscopical diagnosis of AK by a dermatologist, in one or more area(s):

  * Face, ears, (balding) scalp
  * Neck/Shawl area, including the sun-exposed chest area
  * Upper extremities
* Number of AK lesions ≥4 in a continuous treatment area of up to 100 cm2
* AK Olsen grade I-III

Exclusion Criteria:

* Previous field treatment for AK within 2cm of the treatment area, within 3 months
* (non) melanoma skin cancer in treatment area
* Mucosal lesions
* Genetic skin cancer disorder
* Women who are pregnant or breastfeeding
* Women of childbearing potential, who are not willing to use effective contraceptive measures
* Previous allergy or intolerance to either 5FU or calcipotriol
* Patients with known contra-indications for calcipotriol use: previous diagnosis of hyper-calcemia, disturbed calcium metabolism, severe kidney or liver dysfunction
* Concurrent use of oral capecitabine or any other topical or systemic chemopreventive agent for any indication
* Concurrent use of other topical treatments registered as treatment for AK
* Limited understanding of the Dutch language and not being able to give informed consent (incapacitated patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2029-03-02 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Treatment success at 12 months post-treatment | 12 months after finishing treatment
  Treatment success at 12 months post treatment, defined as ≥75% reduction in the number of AK lesions in the treatment area (partial clearance)

SECONDARY OUTCOMES:
AK clearance rate | 3 and 12 months after finishing treatment
  mean percentage change in AK lesions at 3 and 12 months post-treatment
Recurrence rate | 3 and 12 months after finishing treatment
  New lesions and need for retreatment at 3 and 12 months post-treatment
Adverse effects | During treatment and 3 months post-treatment
  Patients experiencing moderate to severe adverse effects
Treatment compliance | During treatment
  Patients who are fully compliant to the prescribed treatment regimen (5FU-CAL or 5FU monotherapy)
Patient satisfaction | 3 and 12 months post-treatment
  Patients who express to be satisfied with their treatment
Quality of life before, during and after treatment | Baseline, 1 week after finishing treatment and 3 and 12 months post-treatment
  The mean score for quality of life on the Skindex-17 questionnaire. The Skindex-17 questionnaire has 17 items investigating the quality of life on different domains. The questions are answered on a five-point scale. A higher score represents a higher impact on QoL.

OTHER OUTCOMES:
Long-term risk for cSCC | at least 3 years post-treatment
  The long-term probability of developing a cSCC

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Zuyderland Medical Center, Heerlen, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg
  - VieCuri Medical Center, Venlo, Limburg
  - Catharina Hospital Eindhoven, Eindhoven, North Brabant

IPD SHARING:
Plan to Share IPD: No